CLINICAL TRIAL: NCT03422588
Title: Intracorporeal Versus Extracorporeal Anastomosis After Laparoscopic Right Colectomy
Brief Title: Surgical Stress and Intracorporeal Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Milone, Professor of Surgery (MD, PhD), Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intrastress-unina
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Laparoscopic Right Colectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal (Experimental): Totally laparoscopic right colectomy with intracorporeal anastomosis
  Interventions: Procedure: Laparoscopic right colectomy
- Extracorporeal (Active Comparator): Laparoscopic assisted right colectomy with extracorporeal anastomosis
  Interventions: Procedure: Laparoscopic right colectomy

INTERVENTIONS:
Procedure: Laparoscopic right colectomy — Laparoscopic right colectomy for colorectal cancer with a standard vascular dissection, performing the anastomosis with a side-to-side mechanical anastomosis fashioned intracorporeally versus extra corporeally

SUMMARY:
The short-term advantages of minimally invasive colon resection have been well established in several randomized trials. A major factor in the development of morbidity is the surgical stress response with subsequent increased demand on the patient's reserves and immune competence. Although the advantage in term of stress response of laparoscopic surgery over open surgery has been widely reported, little is known about the role of Intracorporeal anastomosis.

In an attempt to evaluate the surgical stress response after totally laparoscopic right colectomy a comparative study has been designed.

Two surgical procedures will be evaluated:

* Totally laparoscopic right colectomy with intracorporeal anastomosis (Experimental group)
* Laparoscopic assisted right colectomy with extracorporeal anastomosis (Control group).

ELIGIBILITY:
Inclusion Criteria:

All elective laparoscopic right colectomy for cancer

Exclusion Criteria:

Urgent procedures Immune depressant therapy Immune depressant disease Post-operative Complications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
interleukin 1 | change between time before surgery, 24 hours after surgery, 72 hours after surgery
interleukin 6 | change between time before surgery, 24 hours after surgery, 72 hours after surgery
tumor necrosis factor alpha | change between time before surgery, 24 hours after surgery, 72 hours after surgery
adrenocorticotropic hormone | change between time before surgery, 24 hours after surgery, 72 hours after surgery
cortisol | change between time before surgery, 24 hours after surgery, 72 hours after surgery
insulin | change between time before surgery, 24 hours after surgery, 72 hours after surgery
glucagon | change between time before surgery, 24 hours after surgery, 72 hours after surgery
C-reactive protein | change between time before surgery, 24 hours after surgery, 72 hours after surgery
growth hormone | change between time before surgery, 24 hours after surgery, 72 hours after surgery
prolactin | change between time before surgery, 24 hours after surgery, 72 hours after surgery
fibrinogen | change between time before surgery, 24 hours after surgery, 72 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Milone M, Desiderio A, Velotti N, Manigrasso M, Vertaldi S, Bracale U, D'Ambra M, Servillo G, De Simone G, De Palma FDE, Perruolo G, Raciti GA, Miele C, Beguinot F, De Palma GD. Surgical stress and metabolic response after totally laparoscopic right colectomy. Sci Rep. 2021 May 6;11(1):9652. doi: 10.1038/s41598-021-89183-7. PMID 33958669